CLINICAL TRIAL: NCT01295918
Title: Efficacy of the Probiotic Lactobacillus Reuteri in Prevention of Antibiotic-associated Diarrhea and Clostridium Difficile-related Infections in Hospitalized Children and Adolescents
Brief Title: Probiotic Lactobacillus Reuteri to Prevent Antibiotic-associated Diarrhea and Clostridium Difficile-related Infections in Hospitalized Children
Acronym: AADreuter
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: St Marina University Hospital, Varna, Bulgaria (Other)
Responsible Party: Principal Investigator, Miglena Georgieva, Assoc Prof Miglena Georgieva, MD, PhD, St Marina University Hospital, Varna, Bulgaria., St Marina University Hospital, Varna, Bulgaria
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 128/13.01.2011
Record Dates: First submitted 2011-02-14; First posted 2011-02-15 (Estimated); Last update posted 2013-09-10 (Estimated); Status verified 2013-09

CONDITIONS: Antibiotic Associated Diarrhea; Clostridium Difficile Infection; Gastroenteritis
Keywords: probiotic; AAD; Lactobacillus reuteri; diarrhea
MeSH Terms: conditions — Clostridium Infections; Gastroenteritis; Diarrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo, antibiotic, diarrhea (No Intervention)
- L. reuteri, Antibiotic, diarrhoea (Placebo Comparator): L. reuteri will be ingested by patients on antibiotic therapy, effect of probiotic on AAD will be assessed.
  Interventions: Dietary Supplement: L reuteri in children on antibiotics

INTERVENTIONS:
Dietary Supplement: L reuteri in children on antibiotics — Each patient will be assigned to receive either a probiotic supplement containing 1 x 10 8 CFU Lactobacillus reuteri DSM 17938 in the form of one chewable tablet once per day (BioGaia AB, Stockholm, Sweden) or placebo, identical in taste and appearance. The probiotic or placebo will be taken 2 hours after lunch each day, during the entire period of antibiotic treatment and for an additional 7 days.
  Arms: L. reuteri, Antibiotic, diarrhoea

SUMMARY:
The purpose of this study is to determine if the daily intake of the probiotic Lactobacillus reuteri prevents antibiotic-associated diarrhoea and related Clostridium difficile infections in children and adolescents.

DETAILED DESCRIPTION:
Antibiotic-associated diarrhoea (AAD) occurs in up to 25% of all individuals receiving antibiotics (Bartlett, 2002). In hospitalized patients, AAD is related to significant increases in mortality, length of stay, and cost of medical care (McFarland, 2006). Twenty-nine percent of hospitalized patients may develop diarrhoea after antibiotic use; therefore, identifying strategies to minimize antibiotic-associated diarrhoea could be of significant medical and economic advantage (McFarland, 1998). A promising tool in this area is the probiotic Lactobacillus reuteri

ELIGIBILITY:
Inclusion Criteria:

* 3 - 18 years of age
* Receiving antibiotics for not more than 48 hours prior to enrolment and free from diarrhoea
* The signed informed consent by one/both parents / legal guardian and by the subject if she/he is 12 years or older
* Available throughout the study period
* No use of any other probiotic products during the study period (Bulgarian yoghurt without added probiotics can be used)
* Subject or parents/guardian should have the mental ability to understand and willingness to fulfil all the details of the protocol

Exclusion Criteria:

* Three or more soft and unformed or watery stools per day at admission
* Receiving chemotherapy or radiation therapy
* Diagnosis of inflammatory bowel disease
* Enteral or parenteral nutrition only
* Requiring care in an intensive care unit
* Status post-bowel resection during hospitalization
* Receiving antibiotics four weeks prior to hospitalization
* Patient with severe life threatening illness or immunocompromised (HIV/AIDS, cancer, genetic disorders including cystic fibrosis, children with opportunistic infections, metabolic diseases)
* Pregnancy
* Lack of possibility to store the study product in a temperature below 25°C during the hot season of the year

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2011-02; Primary Completion 2013-06 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
To assess if the probiotic L. reuteri is effective in preventing AAD in children | 2 years
  Incidence of diarrhea during and after treatment with antibiotics in patients ingesting L. reuteri versus placebo during the study period, measured as mean number of episodes per patient. An episode of diarrhea is defined as three or more (≥ 3) soft and unformed or watery bowel movements per day for at least 48 hours.

SECONDARY OUTCOMES:
Incidence of mild diarrhea and severity if diarrhea in children with probiotic treatment | 2 years
  Incidence of mild diarrhoea during and after treatment with antibiotics in patients ingesting L. reuteri versus placebo during the study period is measured as mean number of episodes per patient. An episode of mild diarrhoea is defined as any soft and unformed or watery bowel movements not fulfilling the definition of AAD.
Severity of diarrhoea in patients ingesting L. reuteri versus placebo | 2 years
  Severity of diarrhoea in patients ingesting L. reuteri versus placebo is measured as the total number of soft and unformed or watery bowel movements during an episode of diarrhoea and the presence of blood and mucus in faeces.
Frequency of stool samples positive for C. difficile toxin A and B | 2 years
  Frequency of stool samples positive for C. difficile toxin A and B at baseline, when presenting with diarrhoea during the study period, and at the follow-up 21 days post-antibiotic treatment is done to detect possible clearance of C. difficile, in patients ingesting L. reuteri versus placebo.
Frequencies of other gastrointestinal symptoms | 2 years
  Frequencies of other gastrointestinal symptoms during antibiotic use and 7 and 21 days after cessation of antibiotic use, in the L. reuteri group versus placebo is to be assessed by the validated GSRS score (Gastrointestinal Symptom Rating Score, Svedlund et al., 1988).

CONTACTS AND LOCATIONS:
Overall Officials: Miglena I Georgieva, PhD, Principal Investigator — Pediatric gastroenterology ward
Locations (2):
- Bulgaria (2):
  - St Marina University Hospital, Varna
  - Department of Pediatrics at St Marina University Hospital, Varna, Varna